CLINICAL TRIAL: NCT00832767
Title: Prospective Randomized Controlled Trial of Traditional Laparoscopic Cholecystectomy Versus SILS™ Port Laparoscopic Cholecystectomy
Brief Title: SILS™ Port Laparoscopic Cholecystectomy Post Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS08012
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-05

CONDITIONS: Gallbladder Disease
Keywords: Laparoscopic Cholecystectomy; Single Incision Laparoscopic Surgery; Surgical Procedures, Minimally Invasive
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SILS Port (Active Comparator): SILS™ Port Laparoscopic Cholecystectomy
  Interventions: Procedure: SILS™ port laparoscopic cholecystectomy
- Four Port (Active Comparator): Four Port Laparoscopic Cholecystectomy
  Interventions: Procedure: Four Port Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: SILS™ port laparoscopic cholecystectomy — This interventional arm will have a single incision laparoscopic cholecystectomy procedure.
  Arms: SILS Port
Procedure: Four Port Laparoscopic Cholecystectomy — This interventional arm will have a traditional four port laparoscopic cholecystectomy procedure.
  Arms: Four Port

SUMMARY:
The objectives of this trial are:

1. to assess the feasibility and safety of performing SILS™ Port Laparoscopic Cholecystectomy
2. monitor and compare the outcomes of SILS™ Port Laparoscopic Cholecystectomy versus 4PLC to objectively document the scientific merit and the perceived advantages of SILS™ Port Laparoscopic Cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 85 years old.
* Patient has a diagnosis of biliary colic with documented gallstones or polyps by imaging or Biliary dyskinesia with documented EF < 30%.
* Body Mass Index (BMI) < 45 kg/m2.

Exclusion Criteria:

* Any female patient, who is pregnant, suspected pregnant, or nursing.
* Any patient with acute calculus or acalculous cholecystitis.
* Any patient who has had an upper midline or right sub costal incision.
* Any patient with pre-operative indication for a cholangiogram.
* Any patient with ASA > 3 with normal liver function.
* Any patient who is undergoing Peritoneal Dialysis (PD).
* Any patient who has an unrepaired umbilical hernia or has had prior umbilical hernia repair.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Marks, MD, Principal Investigator — Case Medical Center University Hospitals
Locations (10):
- United States (8):
  - Yale New Haven Medical Center, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - North Shore - Long Island Jewish Health System, Lake Success, New York
  - St. Francis Hospital, Roslyn, New York
  - Case Medical Center, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
- Catholic University of Sacred Heart, Rome, Italy
- Imperial College, England, St. Mary's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Solomon D, Shariff AH, Silasi DA, Duffy AJ, Bell RL, Roberts KE. Transvaginal cholecystectomy versus single-incision laparoscopic cholecystectomy versus four-port laparoscopic cholecystectomy: a prospective cohort study. Surg Endosc. 2012 Oct;26(10):2823-7. doi: 10.1007/s00464-012-2253-0. Epub 2012 May 2. PMID 22549370

RESULTS

PARTICIPANT FLOW:
Groups:
- SILS Port: SILS™ Port Laparoscopic Cholecystectomy
  SILS™ port laparoscopic cholecystectomy : This interventional arm will have a single incision laparoscopic cholecystectomy procedure.
- Four Port: Four Port Laparoscopic Cholecystectomy
  Four Port Laparoscopic Cholecystectomy : This interventional arm will have a traditional four port laparoscopic cholecystectomy procedure.
Period: Overall Study
Arm/Group | SILS Port | Four Port
Started | 121 | 81
Completed | 99 | 63
Not Completed | 22 | 18

BASELINE CHARACTERISTICS:
Population: 202 subjects were enrolled and randomized, however 2 subjects opted not to have surgery and were removed from the study prior to the baseline visit. Therefore data is only available on 200 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | SILS Port | Four Port | Total
Number analyzed (Participants) | 119 | 81 | 200
Age, Customized [Mean (Full Range); unit: years] | 45.8 [18.0 to 77.0] | 44.0 [19.0 to 68.0] | 44.9 [18.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 57 | 148
  Male | 28 | 24 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 7 | 26
  White | 85 | 61 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Safety of SILS™ Port Cholecystectomy Versus 4PLC
Description: Feasibility and safety as determined by intraoperative and postoperative adverse events.
Time Frame: One year
Measure: Number; unit: Participants
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 81
Participants
  At least one AE | 53 | 29
  At least one SAE | 14 | 5
  At least one Device-Related AE or SAE | 6 | 1
  At least one procedure-related AE or SAE | 45 | 23

2. Primary Outcome: Operative Time
Description: Duration of surgical procedure in minutes.
Time Frame: Day 0
Population: One site did not collect the operative time for a patient in the SILS group
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 118 | 81
minutes | 56.8 (23.2) | 45.3 (17.1)

3. Primary Outcome: Estimated Blood Loss
Description: Blood loss from surgical procedure in cc.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 81
cc | 14.9 (35.5) | 14.1 (35.4)

4. Secondary Outcome: Average Pain Experienced in the Last 24 Hours at Various Time Frames
Description: Pain evaluation as determined by a 10-point pain intensity numerical rating scale (PI-NRS) ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Various (Pre-operative, Day 0, 1,3, 5, 1 Week, 2 Week and 1 Month)
Population: Number includes patients who completed pain evaluation questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 81
units on a scale
  Pre-operative | 3.1 (2.7) | 3.3 (2.8)
  Day 0 (Post-operative): number analyzed (Participants) | 117 | 81
  Day 0 (Post-operative) | 6.3 (2.8) | 6.4 (2.3)
  Day 1: number analyzed (Participants) | 118 | 79
  Day 1 | 6.7 (2.5) | 6.1 (2.0)
  Day 3: number analyzed (Participants) | 114 | 79
  Day 3 | 5.4 (2.3) | 4.6 (2.1)
  Day 5: number analyzed (Participants) | 117 | 80
  Day 5 | 4.2 (2.2) | 3.5 (2.1)
  1 Week: number analyzed (Participants) | 116 | 80
  1 Week | 3.5 (2.3) | 2.9 (2.0)
  2 Weeks: number analyzed (Participants) | 115 | 80
  2 Weeks | 2.0 (1.5) | 1.9 (1.5)
  1 Month: number analyzed (Participants) | 113 | 75
  1 Month | 1.8 (1.9) | 1.5 (1.2)

5. Secondary Outcome: Body Image Scale
Description: The Body Image Scale consists of Questions 1-5 on the Body Image Questionnaire. Here, subjects were asked to answer each question on a scale from 1 to 4 with 1 being the best. Therefore, a total score of 5-20 was calculated for each patient with 5 being the best.
Time Frame: Various (1 Week, 2 Week, 1 Month, 3 Month and 1 Year)
Population: The number includes participants who completed the Body Image Questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 116 | 80
units on a scale
  1 Week | 5.6 (1.4) | 5.8 (1.4)
  2 Weeks: number analyzed (Participants) | 115 | 79
  2 Weeks | 5.6 (1.4) | 5.8 (1.4)
  1 Month: number analyzed (Participants) | 114 | 76
  1 Month | 5.5 (1.5) | 5.8 (1.7)
  3 Month: number analyzed (Participants) | 110 | 72
  3 Month | 5.3 (1.0) | 5.5 (1.2)
  1 Year: number analyzed (Participants) | 98 | 62
  1 Year | 5.5 (1.6) | 5.8 (1.9)

6. Secondary Outcome: Cosmetic Scale
Description: The Cosmetic Scale consists of Questions 6-8 on the Body Image Questionnaire. Here, patients were asked to answer questions regarding the cosmesis of their own scar (SILS™) or scars (4PLC). The first 2 questions were answered on a scale from 1 to 7 and Question 8 from 1 to 10, both with 1 being the worst. Therefore, a total score of 3-24 was calculated for each patient with 3 being the worst.
Time Frame: Various (1 Week, 2 Week, 1 Month, 3 Month and 1 Year)
Population: The number includes participants who completed the Cosmetic Scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 116 | 80
units on a scale
  1 Week | 20.5 (3.6) | 18.6 (3.9)
  2 Weeks: number analyzed (Participants) | 115 | 79
  2 Weeks | 21.5 (3.1) | 18.5 (3.9)
  1 Month: number analyzed (Participants) | 114 | 76
  1 Month | 22.1 (2.7) | 19.2 (3.8)
  3 Month: number analyzed (Participants) | 110 | 72
  3 Month | 22.5 (2.6) | 20.0 (3.3)
  1 Year: number analyzed (Participants) | 98 | 62
  1 Year | 22.6 (2.4) | 20.2 (3.7)

7. Secondary Outcome: Confidence Scale Change From Baseline
Description: The Confidence Scale consists of Questions 9 and 10 on the Body Image Questionnaire. One question is before procedure and another is after procedure. The Patients were asked to rate their overall confidence before (baseline) and after the procedure. The scores for before/after procedure range from 1 to 10 with 1 being "not very confident" and 10 being "very confident". The score difference from the before/after treatment is compared between the two procedures (4PLC and SILS™)
  Here, a positive score indicates that patient confidence has increased.
Time Frame: Change from Baseline (Pre-Op) at 1 Week, 2 Week, 1 Month, 3 Month and 1 Year
Population: The number analyzed includes participants who completed questions 9 & 10 on the Body Image Questionnaire. Mean Change from Baseline (Pre-Op).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 116 | 80
units on a scale
  1 Week | 0.5 (2.2) | 0.5 (2.4)
  2 Weeks: number analyzed (Participants) | 115 | 79
  2 Weeks | 0.7 (2.3) | 0.6 (2.2)
  1 Month: number analyzed (Participants) | 114 | 76
  1 Month | 0.5 (2.0) | 0.6 (1.8)
  3 Month: number analyzed (Participants) | 110 | 72
  3 Month | 1.0 (2.3) | 0.6 (1.8)
  1 Year: number analyzed (Participants) | 98 | 62
  1 Year | 1.1 (2.3) | 0.9 (2.7)

8. Secondary Outcome: Normalized Scar Scores
Description: Photo Series Questionnaire (PSQ). All subjects were asked to score their own scar (Question 1), then rate 2 standardized photos (one of 4PLC scars and one of a SILS™ scar) (Questions 2 and 3, respectively) and finally rate their own scar again after viewing the photos (Question 4). All scars were rated on a scale from 1 to 10 with 10 being the best.
  Normalized scores were analyzed for the photo questionnaire. In order to calculate the normalized score, each patient's score of the 4PLC photo was subtracted from their score of their own scar before viewing the photos. the median values were then used to calculate statistical significance.
  Normalized Scores of Own Scar are reported below:
  Question 1 - Question 2 (Q1 - Q2) Question 4 - Question 2 (Q4 - Q2)
  In order to calculate the normalized score for the subject's own scar, Q2 was used as baseline score since Q2 was the score for the conventional procedure 4PLC.
Time Frame: Various (1 Week, 2 Week, 1 Month, 3 Month and 1 Year)
Population: The number includes all participants who completed the Photo Series Questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 81
units on a scale
  Week 1 Q1 - Q2: number analyzed (Participants) | 115 | 80
  Week 1 Q1 - Q2 | 2.8 (2.9) | 0.9 (1.9)
  Week 1 Q4 - Q2: number analyzed (Participants) | 115 | 80
  Week 1 Q4 - Q2 | 3.1 (2.9) | 0.6 (2.0)
  Week 2 Q1 - Q2: number analyzed (Participants) | 115 | 78
  Week 2 Q1 - Q2 | 2.5 (2.5) | 0.4 (1.4)
  Week 2 Q4 - Q2: number analyzed (Participants) | 115 | 78
  Week 2 Q4 - Q2 | 2.7 (2.6) | 0.3 (1.8)
  Month 1 Q1 - Q2: number analyzed (Participants) | 113 | 74
  Month 1 Q1 - Q2 | 2.8 (2.3) | 0.7 (1.5)
  Month 1 Q4 - Q2: number analyzed (Participants) | 113 | 74
  Month 1 Q4 - Q2 | 2.9 (2.3) | 0.2 (1.9)
  Month 3 Q1 - Q2: number analyzed (Participants) | 110 | 72
  Month 3 Q1 - Q2 | 3.0 (2.4) | 0.4 (1.3)
  Month 3 Q4 - Q2: number analyzed (Participants) | 110 | 72
  Month 3 Q4 - Q2 | 3.0 (2.4) | 0.1 (1.3)
  Year 1 Q1 - Q2: number analyzed (Participants) | 98 | 62
  Year 1 Q1 - Q2 | 1.9 (2.0) | -0.0 (1.3)
  Year 1 Q4 - Q2: number analyzed (Participants) | 98 | 62
  Year 1 Q4 - Q2 | 2.0 (1.9) | -0.2 (1.4)

9. Secondary Outcome: Modified Hollander
Description: Surgeons were asked to answer 6 questions regarding the appearance of their subjects' scars. Each patient's score was summed for a total score 0 to 6 with 0 being the best.
Time Frame: Various (1 Week, 2 Week, 1 Month, 3 Month and 1 Year)
Population: The number includes all participants where Modified Hollander Score was completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 115 | 80
units on a scale
  1 Week | 0.37 (0.93) | 0.21 (0.67)
  2 Weeks: number analyzed (Participants) | 114 | 78
  2 Weeks | 0.15 (0.48) | 0.06 (0.29)
  1 Month: number analyzed (Participants) | 112 | 74
  1 Month | 0.10 (0.35) | 0.14 (0.51)
  3 Month: number analyzed (Participants) | 110 | 72
  3 Month | 0.05 (0.27) | 0.01 (0.12)
  1 Year: number analyzed (Participants) | 99 | 63
  1 Year | 0.12 (0.46) | 0.03 (0.18)

10. Secondary Outcome: Physical Quality of Life
Description: SF8 questionnaire was used. This scale measures health and well-being and asks patients to rank their quality of life on a scale of 1 to 5 or a scale of 1 to 6 with 1 being the best and 5 or 6 being the worst. The quality of life questionnaire contains both physical and mental components.
  The raw scores are translated into one from 0 to 100, with 0 representing a very low level of QoL and 100 representing a higher QoL.
Time Frame: Various (Baseline (Pre-Op), Day 1, 3, 5 and 1 Week)
Population: Number includes all participants who completed SF8 Quality of Life Questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 80
units on a scale
  Baseline (Pre-Op) | 49.1 (10.3) | 50.1 (9.2)
  Day 1: number analyzed (Participants) | 118 | 79
  Day 1 | 31.0 (9.9) | 31.8 (8.3)
  Day 3 | 36.8 (9.3) | 40.1 (8.8)
  Day 5: number analyzed (Participants) | 117 | 78
  Day 5 | 42.0 (8.6) | 44.1 (10.6)
  1 Week: number analyzed (Participants) | 117 | 80
  1 Week | 44.4 (9.3) | 47.5 (6.5)

11. Secondary Outcome: Mental Quality of Life
Description: SF8 scale was used. This scale measures health and well-being and asks patients to rank their quality of life on a scale of 1 to 5 or a scale of 1 to 6 with 1 being the best and 5 or 6 being the worst. The quality of life questionnaire contains both physical and mental components.
  The raw scores are translated into one from 0 to 100, with 0 representing a very low level of QoL and 100 representing a higher QoL.
Time Frame: Various (Baseline (Pre-Op), Day 1, 3, 5 and 1 Week)
Population: The number includes participants who completed the SF8 questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 80
units on a scale
  Baseline (Pre-Op) | 47.2 (10.9) | 49.1 (9.4)
  Day 1: number analyzed (Participants) | 118 | 79
  Day 1 | 49.0 (11.2) | 50.6 (9.4)
  Day 3: number analyzed (Participants) | 115 | 80
  Day 3 | 51.4 (8.6) | 51.3 (8.6)
  Day 5: number analyzed (Participants) | 117 | 78
  Day 5 | 52.4 (7.8) | 53.3 (7.4)
  1 Week: number analyzed (Participants) | 117 | 80
  1 Week | 52.0 (8.3) | 53.4 (7.2)

12. Secondary Outcome: Time to Cannulization
Description: Time required to insert SILS port system or 4 individual ports was captured for each procedure in minutes.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SILS Port | Four Port
Number analyzed (Participants) | 119 | 81
minutes | 6.3 (4.4) | 6.9 (3.9)

ADVERSE EVENTS:
Time Frame: AEs collected from enrollment through end of study which was a period of 1 year.
Arm/Group | SILS Port | Four Port
Serious Adverse Events (participants affected / at risk) | 15/119 | 5/81
Other Adverse Events (participants affected / at risk) | 44/119 | 27/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SILS Port (N=119) | Four Port (N=81)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Incisional hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 1 (3) | 0 (0)
Urinary Retention Postoperative (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Urinary Tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SILS Port (N=119) | Four Port (N=81)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 6 (6)
Nausea (Gastrointestinal disorders) | 11 (12) | 6 (7)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7)
Abdominal Pain (Gastrointestinal disorders) | 14 (15) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No